CLINICAL TRIAL: NCT01000233
Title: Value of Oral Phytate (InsP6) in the Prevention of Progression of the Cardiovascular Calcifications
Acronym: CALCIFICA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Laboratorios BIOMED SA (Unknown)
Responsible Party: Carlos Fernandez-Palomeque, Hospital Universitari Son Dureta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIS_PI081931
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Heart Valve Disease; Aortic Stenosis
Keywords: PATOLOGIC CALCIFICATION; AORTIC VALVE STENOSIS; INOSITOL HEXAPHOSPHATE
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis | interventions — Phytic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phytine (Phytate) (Active Comparator): 300 mg tid* 24 months
  Interventions: Dietary Supplement: Phytine (phytate); Dietary Supplement: Placebo
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phytine (phytate) — 300 mg tid * 24 months
  Other Names: LITSTOP; Inositol hexaphosphate
  Arms: Phytine (Phytate)
Dietary Supplement: Placebo — Phytine (Phytate)
  Other Names: LITSTOP; Inositol hexaphosphate

SUMMARY:
Intervention study focused on preventing the progression of aortic valve calcification.

Vascular and cardiac calcifications are a marker of risk and poor outcome, especially the severe calcified aortic stenosis and coronary calcification.

Its increasing prevalence is now a health problem. The knowledge and the therapeutic objective of this condition have changed in recent years and pathophysiological aspects at present, focus on atherosclerotic disease and inflammation.

Several clinical trials have failed to demonstrate that statins or ACE inhibitors prevent the progression of cardiovascular calcification.

Taking into account the new concepts of ectopic calcification and research results from our group, the most logical approach to prevent progression would be an early intervention and management of the calcification inhibiting agents such as phytate (inositol six-phosphate -- InsP6).

Hypothesis: The phytate prevents or delays the progression of cardiovascular calcification.

It is a clinical trial of intervention of oral phytate (InsP6) in patients with mild to moderate cardiovascular calcification (aortic valve and / or coronary arteries) compared with placebo over a period of 24 months.

It is a prospective, randomized minimization of variables to ensure homogeneity of the groups.

The primary analysis will be the time evolution of the extent of calcium in the aortic valve and coronary arteries made with CT.

Secondary variables are the degree of progression of aortic stenosis and clinical events (death, stroke, angina, stroke and cancer of any type).

DETAILED DESCRIPTION:
Main objective of the study:

To evaluate whether the progression of aortic valve calcification and/or coronary arteries in the group treated with oral InsP6 is smaller than in the placebo group, measured by quantification of calcium (score and mass) by multidetector CT to the inclusion in the study and 24 months.

Secondary:

To observe whether the progression of aortic stenosis severity in the intervention group is smaller than in the placebo group, evaluated by echocardiography.

To compare the clinical events between the intervention and placebo groups, measured as the combined event of death, hospitalization for angina, coronary revascularization (surgical or percutaneous), nonfatal myocardial infarction and stroke of any type.

To compare the adverse effects collected by spontaneous reporting between the two groups.

Main variable of analysis ( multidetector CT measurements): Calcium in aortic valve and/or coronary arteries assessed by Agatston units (AU) on two occasions: before treatment, and 2 years of follow up.

Types of analysis of the main variable:

* Percentage of change in quantity of calcium in aortic valve between baseline and study end.
* Absolute difference from quantity of calcium in aortic valve between baseline and study end.
* Percentage change in coronary calcium quantity between baseline and study end.
* Absolute difference in coronary calcium quantity between baseline and study end.
* Percentage change of total calcium in aortic valve and coronary artery between baseline and study end.
* Absolute difference of total calcium in aortic valve and coronary artery between baseline and study end.

Secondary analysis:

Progression of aortic stenosis severity assessed by gradient and maximum speed, average by echocardiography.

Percentage of clinical events. The event is considered the composite event "death, hospitalization for angina, coronary revascularization (surgical or percutaneous), valvular surgery, nonfatal myocardial infarction or stroke of any type"

Measurements:

Calcium valve by echocardiography: expressed as Rosenhek score at the aortic and coronary calcium CT MD: expressed as Agatston score units and mass determination of calcium. Measurement of emitted radiation .

Demographic variables: age, sex, race, weight, height, and BMI SC, snuff and alcohol habits.

Food Survey: Quality and frequency of feeding in relation to income Ins6P. Conventional hematological and biochemical parameters: blood count. ESR. Urea, Creatinine, Na, K, Ca, P Phytate: determination in urine by InsP6 technique developed at the Universitat Illes Balears. The blind is maintained until final results.

Events qualifiers: death, nonfatal myocardial infarction, hospitalization for angina, coronary revascularization, stroke (score by Events Committee of the study).

Adverse events: Determination of adverse events according to RD 223/2004 (Spanish regulation) Patient Compliance: By counting returned capsules and quantification of phytate in urine.

Withdrawals: If there are withdrawals for any reason the patient is requested authorization for calcium measurement by CT when possible.

Statistical:

Predetermination of sample size:

Assuming the evolution of aortic valve calcification between 21.7% to 32% per year found in the placebo arm of clinical trials with similar methodology and population, and based on a standard deviation of 1100 AU per year, assuming a Type I error of 0.05 and type II of 0.2, to detect a difference of 20% annually between treatments, we need between 124 and 105 patients, respectively, assuming a 10% of losses, and an average Agatston units at baseline, of 1700. We decide to adopt the larger size.

Strategy for statistical analysis: The analysis of data will carry out maintaining the blind and conducted by intention to treat and, as a secondary analysis, per protocol.

The population for the intention to treat analysis, include those randomized patients who have received at least one dose of assigned treatment. The per protocol population will consist of those individuals who finish the study without protocol violation.

A description of the baseline characteristics of the groups, will be carry out, verifying, despite using a system of random assignment, the homogeneity of the two groups for baseline variables. A test for the normality of quantitative variables to select the statistic descriptors, mean (CI95%) or median (RI), and test for comparisons.

The main result will be a change of aortic valve calcification, calculated as the percentage change from baseline divided by the duration of follow up as years. An analysis stratified for each independent variable.

An increment of at least 18% of the basal calcification, will be considered evident progression, by contrast, a lesser progression will be considered response to treatment. Logistic regression will be used to establish the likelihood of response.

Secondary objectives will be analyzed by comparing the ratios between treatment groups.

There will be a descriptive analysis of the side effects listed in both groups.

Ethical considerations: No special ethical problems arise in the trial because of the phytate is considered a safe product (FDA-Title 21 subchapter GRSH E-Part 582) which are a component of the normal diet, and because of the chances of problems with excessive intake of this are nil. Nor is amended nor intervene during the study in routine clinical practice.

The most important aspect is to control the radiation dose that patients receive during the multidetector CT. In any case is lower than the environmental background radiation received during 6 months.

Considering this aspect, intermediate CT study has not been scheduled.

No information is available on the extent of calcium through multidetector-CT to let us build the sample size with great confidence. We have used the values of progressive studies Cowell and Houslay for making this approximation.

ELIGIBILITY:
Inclusion Criteria:

* Calcium in the aortic valve, characterized by Rosenhek score grade 2 or 3 in echocardiography and / or with not severe coronary calcification detected in other studies (angiography, CT).

Exclusion criteria:

* Severe aortic (Rosenhek 4)or coronary calcification .
* Positive pregnancy test (if pregnancy occurs during the study be deferred final evaluation at the end of gestation, if the patient wishes to continue in the study).
* Addiction to drugs or alcohol.
* Renal insufficiency (serum creatinine> 2mg/dl).
* Liver disease or cirrhosis.
* Severe valve disease or requiring surgery during the study.
* Unstable ischemic heart disease (revascularization in the last 3 months).
* Atrial fibrillation in the initial evaluation (difficulty in measuring Ca). May be included later if sinus rhythm is achieved stable for at least three months.
* The need for any medication in relation to calcium metabolism (PTH, bisphosphonates, strontium ranelate, raloxifene, oral calcium, vitamin D, calcitonin, etc.).
* Participation in another trial in the three months prior to evaluation.
* Suspected difficulties to accomplish during the two years, for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-03 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Calcium in aortic valve and in coronary arteries assessed by multidetector CT scanner (Agatston units) | 24 months

SECONDARY OUTCOMES:
Clinical events. A composite event is considered: death, hospitalization for angina, coronary revascularization (surgical or percutaneous), valvular surgery, nonfatal myocardial infarction and stroke. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Frontera, MD, Study Chair — Hospital Universitario Son Dureta
Locations (1):
- Hospital Universitario Son Dureta, Palma, Balearic Islands, Spain

REFERENCES:
- [Background] Grases F, Prieto RM, Simonet BM, March JG. Phytate prevents tissue calcifications in female rats. Biofactors. 2000;11(3):171-7. doi: 10.1002/biof.5520110303. PMID 10875304
- [Background] Grases F, Sanchis P, Perello J, Isern B, Prieto RM, Fernandez-Palomeque C, Saus C. Phytate reduces age-related cardiovascular calcification. Front Biosci. 2008 May 1;13:7115-22. doi: 10.2741/3214. PMID 18508720
- [Background] Grases F, Sanchis P, Costa-Bauza A, Bonnin O, Isern B, Perello J, Prieto RM. Phytate inhibits bovine pericardium calcification in vitro. Cardiovasc Pathol. 2008 May-Jun;17(3):139-45. doi: 10.1016/j.carpath.2007.08.005. Epub 2007 Oct 24. PMID 18402805
- [Background] Grases F, Sanchis P, Perello J, Isern B, Prieto RM, Fernandez-Palomeque C, Torres JJ. Effect of crystallization inhibitors on vascular calcifications induced by vitamin D: a pilot study in Sprague-Dawley rats. Circ J. 2007 Jul;71(7):1152-6. doi: 10.1253/circj.71.1152. PMID 17587727